CLINICAL TRIAL: NCT02544750
Title: A Double-blind, Randomized, Placebo-controlled Study to Investigate the Efficacy and Safety of Cannabidiol (GWP42003-P, CBD) as Add-on Therapy in Patients With Tuberous Sclerosis Complex Who Experience Inadequately-controlled Seizures
Brief Title: An Open-label Extension Trial of Cannabidiol (GWP42003-P, CBD) for Seizures in Tuberous Sclerosis Complex (GWPCARE6)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: GW Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWEP1521 Open-Label Extension; 2015-002154-12 (EudraCT Number)
Record Dates: First submitted 2015-09-07; First posted 2015-09-09 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Tuberous Sclerosis Complex; Seizures
MeSH Terms: conditions — Tuberous Sclerosis; Seizures | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GWP42003-P (Experimental): 100 mg/mL GWP42003-P oral solution taken twice daily (morning and evening). Participants will be dosed up to a maximum of 50 mg/kg/day. Dose may be lower if Investigator judges benefit and/or tolerability issues.
  Interventions: Drug: GWP42003-P

INTERVENTIONS:
Drug: GWP42003-P — Yellow oily solution containing cannabidiol dissolved in the excipients sesame oil and anhydrous ethanol with added sweetener (sucralose) and strawberry flavoring.
  Other Names: Cannabidiol; CBD

SUMMARY:
This trial consists of 2 parts: a double-blinded phase and an open-label extension phase. The open-label extension phase only will be described in this record. All participants will receive the same dose of GWP42003-P. However, investigators may subsequently decrease or increase the participant's dose until the optimal dose is found.

ELIGIBILITY:
Key Inclusion Criteria:

* Completion of the GWEP1521 Blinded Phase

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thiele EA, Bebin EM, Bhathal H, Jansen FE, Kotulska K, Lawson JA, O'Callaghan FJ, Wong M, Sahebkar F, Checketts D, Knappertz V; GWPCARE6 Study Group. Add-on Cannabidiol Treatment for Drug-Resistant Seizures in Tuberous Sclerosis Complex: A Placebo-Controlled Randomized Clinical Trial. JAMA Neurol. 2021 Mar 1;78(3):285-292. doi: 10.1001/jamaneurol.2020.4607. PMID 33346789
- [Result] Thiele EA, Bebin EM, Filloux F, Kwan P, Loftus R, Sahebkar F, Sparagana S, Wheless J. Long-term cannabidiol treatment for seizures in patients with tuberous sclerosis complex: An open-label extension trial. Epilepsia. 2022 Feb;63(2):426-439. doi: 10.1111/epi.17150. Epub 2021 Dec 27. PMID 34957550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 199 participants with tuberous sclerosis complex (TSC) who met all inclusion criteria and no exclusion criteria and completed the double-blind study GWEP1521 (NCT02544763) were enrolled into this Open-label Extension (OLE) study to receive GWP42003-P.
Pre-assignment Details: OLE investigational medicinal product (IMP) was titrated up to 25 mg/kg/day while blinded IMP was simultaneously tapered down to zero to accommodate those participants who had been randomized to placebo during the double-blind phase (DBP) of the study. All participants were to complete the transition and enter the OLE taking 25 mg/kg/day GWP42003-P.
Groups:
- GWP42003-P (Double-blind Phase): Participants who had received GWP42003-P during the double-blind phase and then GWP42003-P in the OLE phase.
- Placebo (Double-blind Phase): Participants who had received placebo during the double-blind phase and then GWP42003-P in the OLE phase.
Period: Overall Study
Arm/Group | GWP42003-P (Double-blind Phase) | Placebo (Double-blind Phase)
Started | 124 | 75
Completed | 22 | 12
Not Completed | 102 | 63
Not completed — Physician Decision | 3 | 1
Not completed — Other reasons | 69 | 39
Not completed — Met withdrawal criteria | 2 | 2
Not completed — Transition To Commercial Product | 1 | 0
Not completed — Withdrawal by Parent/Guardian | 8 | 7
Not completed — Adverse Event | 8 | 10
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GWP42003-P (Double-blind Phase) | Placebo (Double-blind Phase) | Total
Number analyzed (Participants) | 124 | 75 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.69 (9.64) | 13.92 (10.63) | 13.15 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 30 | 81
  Male | 73 | 45 | 118
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 111 | 66 | 177
  Black/African American | 4 | 0 | 4
  American Indian/Alaska Native | 1 | 0 | 1
  Asian | 1 | 3 | 4
  Other | 7 | 6 | 13
Baseline Tuberous Sclerosis Complex (TSC)-Associated Seizures [Median (Full Range); unit: Seizures] — TSC-associated seizures included: focal motor seizures without impairment of consciousness or awareness (Type 1 focal motor); focal seizures with impairment of consciousness or awareness (Type 2 focal); focal seizures evolving to bilateral generalized convulsive seizures (Type 3 focal); and tonic clonic, tonic, clonic, or atonic seizures that are countable. The Baseline Period included all data prior to Day 1. Population: Seizure frequency was assessed in the OLE Safety Analysis Set.
  Seizures | 58.08 [7.7 to 432.0] | 55.10 [8.0 to 558.0] | 56.90 [7.7 to 558.0]
Baseline Total Seizures [Median (Full Range); unit: Seizures] — Total seizures included all seizure types combined. The Baseline Period included all data prior to Day 1. Population: OLE Safety Analysis Set
  Seizures | 59.95 [7.7 to 595.0] | 56.97 [8.0 to 1660.1] | 58.90 [7.7 to 1660.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events, Discontinuations Due to AEs, Serious AEs, and Treatment-related AEs (TEAE)
Description: An adverse event (AE) was defined as any new unfavorable/unintended signs/symptoms (including abnormal laboratory findings), or diagnosis or worsening of a pre-existing condition, which occurred following screening and at any point up to the post-treatment safety follow-up visit, which may or may not be related to the IMP. An AE that started, or worsened in severity or seriousness, following the first dose of IMP was considered a TEAE. A serious AE was defined as any AE that results in any of the following outcomes: death, life-threatening adverse experience, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or cancer, any other experience that suggests a significant hazard, contraindication, side effect or precaution that may require medical or surgical intervention to prevent one of the outcomes listed above, or an event that changes the risk/benefit ratio of the study.
Time Frame: OLE Day 1 up to 4 years
Population: Adverse events were assessed in the OLE Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Double-blind Phase): Participants who had received placebo during double-blind phase and then GWP42003-P in the OLE phase.
Arm/Group | GWP42003-P (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 124 | 75
Participants
  Any TEAE | 117 | 75
  Any treatment-related TEAE | 80 | 60
  Any TEAE leading to permanent discontinuation of IMP | 11 | 7
  Any treatment-related TEAE leading to permanent discontinuation of IMP | 9 | 7
  Any serious TEAE | 38 | 18
  Any treatment-related serious TEAE | 7 | 8
  Any fatal TEAEs | 1 | 0

2. Primary Outcome: Number of Participants With Any TEAE, by Severity
Description: An adverse event (AE) was defined as any new unfavorable/unintended signs/symptoms (including abnormal laboratory findings), or diagnosis or worsening of a pre-existing condition, which occurred following screening and at any point up to the post-treatment safety follow-up visit, which may or may not be related to the IMP. An AE that started, or worsened in severity or seriousness, following the first dose of IMP was considered a TEAE.
  Grade 1 (Mild) is defined as asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 (Moderate) is defined as minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental activities of daily living (ADL). Grade 3 (Severe) is defined as medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
Time Frame: OLE Day 1 up to 4 years
Population: Adverse events were assessed in the OLE Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 124 | 75
Participants
  Mild TEAE | 35 | 16
  Moderate TEAE | 63 | 48
  Severe TEAE | 19 | 11

3. Secondary Outcome: Percent Change From Baseline in the Number of TSC-associated Seizures During the OLE Treatment Period
Description: TSC-associated seizures include: focal motor seizures without impairment of consciousness or awareness; focal seizures with impairment of consciousness or awareness; focal seizures evolving to bilateral generalized convulsive seizures and tonic-clonic, tonic, clonic or atonic seizures. A negative percent change from baseline indicates improvement.
Time Frame: OLE Day 1 up to 4 years
Population: TSC-associated seizures were assessed in the OLE Safety Analysis Set.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | GWP42003-P (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 124 | 75
percent change | -55.66 [-86.47 to -12.33] | -46.76 [-78.17 to -15.69]

4. Secondary Outcome: Number of Participants Considered Treatment Responders During the OLE Treatment Period
Description: Treatment responders were defined as those participants with a ≥50% reduction from baseline in TSC-associated seizure frequency, during the treatment period, for participants who had not withdrawn from the trial during the treatment period. TSC-associated seizures included: focal motor seizures without impairment of consciousness or awareness (Type 1 focal motor); focal seizures with impairment of consciousness or awareness (Type 2 focal); focal seizures evolving to bilateral generalized convulsive seizures (Type 3 focal); and tonic-clonic, tonic, clonic, or atonic seizures that were countable. Participants who withdrew from the trial during the treatment period were considered non-responders.
Time Frame: OLE Day 1 up to 4 years
Population: Treatment responders were assessed in the OLE Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 124 | 75
Participants
  ≥ 50% reduction: Yes | 70 | 36
  ≥ 50% reduction: No | 54 | 39

5. Secondary Outcome: Caregiver Global Impression of Change (CGIC) and Subject Global Impression of Change (SGIC) Score During the OLE Treatment Period
Description: The CGIC comprised the following question to be rated on a 7-point scale (1, Very Much Improved; 2, Much Improved; 3, Slightly Improved; 4, No Change; 5, Slightly Worse; 6, Much Worse; 7, Very Much Worse): "Since your child started treatment, please assess the status of your child's overall condition (comparing their condition now to their condition before treatment)." The SGIC comprised the following question to be rated on a 7-point scale (1, Very Much Improved; 2, Much Improved; 3, Slightly Improved; 4, No Change; 5, Slightly Worse; 6, Much Worse; 7, Very Much Worse): "Since you started treatment, please assess the status of your overall condition (comparing your condition now to your condition before treatment)." The average CGIC and SGIC scores are being reported, with higher values indicating worse condition.
Time Frame: OLE Day 1 and up to 4 years
Population: Caregiver Global Impression of Change and Subject Global Impression of Change were assessed in the OLE Safety Analysis Set in participants with available data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003-P (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 40 | 28
score on a scale
  Caregiver: number analyzed (Participants) | 39 | 25
  Caregiver | 3.2 (1.58) | 3.4 (1.12)
  Subjects: number analyzed (Participants) | 3 | 3
  Subjects | 4.0 (0.0) | 2.7 (1.53)
  Combined Caregiver and Subjects | 3.2 (1.56) | 3.3 (1.16)

6. Secondary Outcome: Percent Change From Baseline in Total Seizure Frequency During the OLE Treatment Period
Description: Total seizures included all seizure types, eg. combination of TSC-associated and other seizures. TSC-associated seizures included: focal motor seizures without impairment of consciousness or awareness (Type 1 focal motor); focal seizures with impairment of consciousness or awareness (Type 2 focal); focal seizures evolving to bilateral generalized convulsive seizures (Type 3 focal); and tonic-clonic, tonic, clonic, or atonic seizures that were countable. A negative percent change from baseline indicates improvement in total seizure frequency.
Time Frame: OLE Day 1 up to 4 years
Population: Total seizure frequency was assessed in the OLE Safety Analysis Set.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | GWP42003-P (Double-blind Phase) | Placebo (Double-blind Phase)
Number analyzed (Participants) | 124 | 75
percent change | -55.18 [-84.21 to -11.95] | -46.76 [-76.22 to -19.77]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from OLE Day 1 up to 4 years.
Description: An adverse event (AE) was defined as any new unfavorable/unintended signs/symptoms (including abnormal laboratory findings), or diagnosis or worsening of a pre-existing condition, which occurred following screening and at any point up to the post-treatment safety follow-up visit, which may or may not be related to the IMP. TEAEs were defined as AEs with a start date on or after the first dose of IMP in the OLE Day 1.
Arm/Group | Placebo (Double-blind Phase) | GWP42003-P (Double-blind Phase)
All-Cause Mortality (participants affected / at risk) | 1/124 | 0/75
Serious Adverse Events (participants affected / at risk) | 38/124 | 18/75
Other Adverse Events (participants affected / at risk) | 117/124 | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Phase) (N=124) | GWP42003-P (Double-blind Phase) (N=75)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Soft tissue inflammation (General disorders) | 1 | 0
Adenoiditis (Infections and infestations) | 1 | 0
Adenovirus infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Enterovirus infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis astroviral (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Implant site infection (Infections and infestations) | 1 | 0
Infective myositis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 5 | 0
Laryngitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Anticonvulsant drug level increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Astrovirus test positive (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 1
Influenza A virus test positive (Investigations) | 1 | 0
Investigation (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Liver function test increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Respiratory syncytial virus test positive (Investigations) | 1 | 0
Sapovirus test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 2
Weight decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Fluid intake reduced (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Kidney angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Change in seizure presentation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epileptic encephalopathy (Nervous system disorders) | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 0
Postictal state (Nervous system disorders) | 1 | 0
Sedation (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 12 | 4
Seizure cluster (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 9 | 1
Syncope (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alcohol use (Social circumstances) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Double-blind Phase) (N=124) | GWP42003-P (Double-blind Phase) (N=75)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 12 | 9
Diarrhoea (Gastrointestinal disorders) | 50 | 43
Nausea (Gastrointestinal disorders) | 3 | 4
Retching (Gastrointestinal disorders) | 3 | 3
Vomiting (Gastrointestinal disorders) | 27 | 13
Fatigue (General disorders) | 7 | 10
Pyrexia (General disorders) | 33 | 15
Bronchitis (Infections and infestations) | 2 | 5
Conjunctivitis (Infections and infestations) | 8 | 3
Ear infection (Infections and infestations) | 6 | 3
Gastroenteritis (Infections and infestations) | 5 | 2
Gastroenteritis viral (Infections and infestations) | 7 | 3
Influenza (Infections and infestations) | 16 | 4
Nasopharyngitis (Infections and infestations) | 19 | 16
Otitis media (Infections and infestations) | 8 | 4
Pharyngitis (Infections and infestations) | 8 | 2
Pharyngitis streptococcal (Infections and infestations) | 13 | 4
Pneumonia (Infections and infestations) | 5 | 3
Rhinitis (Infections and infestations) | 4 | 1
Sinusitis (Infections and infestations) | 7 | 2
Upper respiratory tract infection (Infections and infestations) | 22 | 10
Urinary tract infection (Infections and infestations) | 7 | 3
Viral infection (Infections and infestations) | 4 | 5
Viral upper respiratory tract infection (Infections and infestations) | 4 | 3
Accident (Injury, poisoning and procedural complications) | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 6 | 4
Fall (Injury, poisoning and procedural complications) | 13 | 8
Head injury (Injury, poisoning and procedural complications) | 4 | 0
Laceration (Injury, poisoning and procedural complications) | 9 | 4
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 3
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 3
Tooth fracture (Injury, poisoning and procedural complications) | 5 | 1
Alanine aminotransferase increased (Investigations) | 8 | 6
Aspartate aminotransferase increased (Investigations) | 6 | 4
Blood prolactin increased (Investigations) | 2 | 3
Gamma-glutamyltransferase increased (Investigations) | 4 | 9
Liver function test increased (Investigations) | 2 | 6
Weight decreased (Investigations) | 7 | 9
Weight increased (Investigations) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 23 | 24
Ataxia (Nervous system disorders) | 4 | 5
Dizziness (Nervous system disorders) | 5 | 4
Generalised tonic-clonic seizure (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 9 | 5
Lethargy (Nervous system disorders) | 3 | 5
Sedation (Nervous system disorders) | 2 | 4
Seizure (Nervous system disorders) | 40 | 19
Somnolence (Nervous system disorders) | 15 | 24
Abnormal behaviour (Psychiatric disorders) | 6 | 5
Aggression (Psychiatric disorders) | 5 | 9
Agitation (Psychiatric disorders) | 7 | 2
Anxiety (Psychiatric disorders) | 4 | 3
Insomnia (Psychiatric disorders) | 5 | 6
Intentional self-injury (Psychiatric disorders) | 4 | 0
Irritability (Psychiatric disorders) | 9 | 5
Sleep disorder (Psychiatric disorders) | 6 | 4
Urinary retention (Renal and urinary disorders) | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1
Toothache (Gastrointestinal disorders) | 4 | 0
Gait disturbance (General disorders) | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 4
Status epilepticus (Nervous system disorders) | 9 | 1
Mental status changes (Psychiatric disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT02544750/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT02544750/SAP_001.pdf